CLINICAL TRIAL: NCT02888509
Title: Neural and Cognitive Mechanisms of Depression and Anxiety: a Multimodal MRI Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, chenhuafu, professor, University of Electronic Science and Technology of China
Other Study IDs: UESTC-chenhuafulab-002
Record Dates: First submitted 2016-08-30; First posted 2016-09-05 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-08

CONDITIONS: Depression
Keywords: depression; anxiety disorder; bipolar disorder; Magnetic Resonance Imaging
MeSH Terms: conditions — Depression; Anxiety Disorders; Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- healthy control: Well mathed with patients in age, gender, education
- major depression disorder: patients with major depression disorder
- anxiety disorder: patients with anxiety disorder
- bipolar depression disorder: patients with bilopar depression disorder

SUMMARY:
To explore the neural and cognitive mechanisms of depression (including unipolar depression and Bipolar disorder) and anxiety using multimodal MRI techniques.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 16 to 55 years old.
* All patients were interviewed by two experienced psychiatrists using the Structured Clinical Interview for DSM-IV (patient edition)

Exclusion Criteria:

* Schizophrenia, mental retardation or personality disorder, any history of loss of consciousness, substance abuse, serious medical or neurological illness.
* Subjects with contraindications to MRI

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with major depression, bilopar, anxiety disorders were recruited from the mental health center of Chengdu, Sichuan, China.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Brain structural and functional changes in patients | one time point
  Structure and function changes in patients will be assessed by Voxel-based morphometry analysis for structural changes, as well as Regional homogeneity, Amplitude of lowfrequency fluctuation, etc, for functional changes.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Life Science and Technology, University of Electronic Science and Technology, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen Y, Cui Q, Sheng W, Tang Q, Lu F, Pang Y, Nan X, He Z, Li D, Lei T, Chen H. Anomalous neurovascular coupling in patients with generalized anxiety disorder evaluated by combining cerebral blood flow and functional connectivity strength. Prog Neuropsychopharmacol Biol Psychiatry. 2021 Dec 20;111:110379. doi: 10.1016/j.pnpbp.2021.110379. Epub 2021 Jun 7. PMID 34111495
- [Derived] Yang Y, Cui Q, Pang Y, Chen Y, Tang Q, Guo X, Han S, Ameen Fateh A, Lu F, He Z, Huang J, Xie A, Li D, Lei T, Wang Y, Chen H. Frequency-specific alteration of functional connectivity density in bipolar disorder depression. Prog Neuropsychopharmacol Biol Psychiatry. 2021 Jan 10;104:110026. doi: 10.1016/j.pnpbp.2020.110026. Epub 2020 Jul 2. PMID 32621959
- [Derived] Wang Y, Wang X, Ye L, Yang Q, Cui Q, He Z, Li L, Yang X, Zou Q, Yang P, Liu D, Chen H. Spatial complexity of brain signal is altered in patients with generalized anxiety disorder. J Affect Disord. 2019 Mar 1;246:387-393. doi: 10.1016/j.jad.2018.12.107. Epub 2018 Dec 26. PMID 30597300